CLINICAL TRIAL: NCT03672604
Title: A Phase 1, Single- and Multiple-Dose, Double-Blind, Randomized, Placebo-Controlled, Dose-Escalating Study to Assess the Safety, Tolerability, and Pharmacokinetics of NLY01 in Healthy Subjects
Brief Title: A Phase 1 Study to Assess the Safety of NLY01 in Healthy Subjects
Acronym: NLY01-H1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuraly, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-NRALY-PHAS1-M-0000
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Safety and Tolerability in Healthy Volunteers
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: A Phase 1, first-in-human, double-blind, randomized, placebo-controlled, single-ascending followed by multiple-dose study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Single Dose (Placebo Comparator): Cohort 1 = 0.25 mg NLY01 Cohort 2 = 0.8 mg NLY01 Cohort 3 = 2.5 mg NLY01 Cohort 4 = 5 mg NLY01 Cohort 5 = 10 mg NLY01
  All cohorts include 8 subjects randomized to receive a single dose of NLY01 or placebo (6 active, 2 placebo).
  Interventions: Drug: NLY01
- Part B: Multiple Dose (Placebo Comparator): In Part B, NLY01 or placebo will be administered once-weekly for 4 doses. There will be 3 sequentially-enrolled, ascending-dose cohorts of 8 subjects (6 active, 2 placebo). Doses in Part B will be a fraction of the maximum tolerated dose (MTD) established in Part A.
  Cohort 6 = 15% of the single-dose MTD Cohort 7 = 35% of the single-dose MTD Cohort 8 = 70% of the single-dose MTD
  Interventions: Drug: NLY01
- Part C:Multiple Dose (Placebo Comparator): In Part C, NLY01 or placebo will be administered once-weekly for 6 doses.
  Cohort 10 = 2.5 mg NLY01 Cohort 11 = 5 mg NLY01
  Interventions: Drug: NLY01

INTERVENTIONS:
Drug: NLY01 — NLY01, a PEGylated form of the anti-diabetic peptide exenatide
  Other Names: Placebo; normal saline

SUMMARY:
This is a Phase 1, first-in-human study designed to assess the safety, tolerability, and pharmacokinetics of NLY01, a PEGylated form of exenatide, in healthy volunteers. NLY01 is being developed as a potential treatment for neurodegenerative disorders including Parkinson's disease. This study is intended to identify the appropriate dose-range for evaluation in Parkinson's disease patients.

DETAILED DESCRIPTION:
This is a Phase 1, first-in-human, double-blind, randomized, placebo-controlled, single and multiple-dose study to assess the safety, tolerability, and PK of NLY01, a PEGylated form of the anti-diabetic peptide exenatide, when administered by SC injection in healthy subjects.

In Part A of the study, 5 ascending-dose cohorts will be sequentially enrolled with an evaluation of safety and tolerability prior to each dose-escalation. Subjects in each cohort will be randomized to receive NLY01 or placebo. Each dose escalation and selection of doses for Part B will be conducted with oversight by an independently-chaired Safety Review Committee.

In Part B, subjects will receive once-weekly subcutaneous doses of NLY01 or placebo for 4 weeks. Three ascending-dose cohorts will be sequentially-enrolled with a safety review prior to each dose-escalation. Subjects in all Part B cohorts will receive fixed doses of NLY01 (or placebo) once-weekly for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18 to 65 years of age, inclusive.
* BMI ≥ 18.5 and ≤ 32.0 kg/m2 at screening and check-in. BMI = weight (kg)/(height [m])2.
* Women of child-bearing potential must agree to use a medically acceptable method of contraception from screening through 30 days after the final dose of study drug.
* Non-childbearing potential.
* Men who are sexually active and whose partners are women of child-bearing potential must agree to use condoms from screening through 90 days after administration of study drug, and their partners must be willing to use a medically acceptable method of contraception (a barrier method, intrauterine device, or hormonal contraception) from screening through 90 days after administration of the last dose of study drug.
* Men must agree to not donate sperm from screening through 90 days after study drug administration.
* Subjects must be able to communicate effectively with the study personnel.
* Subjects must be healthy and without clinically significant abnormalities as assessed by review of medical and surgical history, physical examination, vital signs measurement, ECG, and laboratory evaluations conducted at screening and on Day -1 Check-in. A single repeat measurement/test may be performed to confirm vital signs, ECG, and clinical laboratory tests abnormalities (ie, to confirm that a subject is eligible).
* Subjects must be nonsmokers, defined as having abstained from tobacco- or nicotine containing products (eg, cigarettes, chewing tobacco, snuff, nicotine patches, and electronic cigarettes) in the 6 months prior to screening.
* Subjects must be informed of the nature and risks of the study and give written informed consent prior to screening.

Exclusion Criteria:

* Positive pregnancy test or is lactating/breastfeeding.
* History or presence of conditions which, in the judgment of the investigator, are known to interfere with the distribution, metabolism, or excretion of drugs.
* History or presence of conditions that may place the subject at increased risk as determined by the investigator.
* History of surgery or major trauma within 12 weeks of screening, or surgery planned during the study.
* History of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction within 12 months of screening.
* Use of prescription, OTC drugs (including herbal preparations) within 7 days or 5 half lives (if known), whichever is longer, prior to administration of the first dose of study drug.
* Has received a vaccination within 14 days prior to administration of the first dose of study drug.
* Has taken other investigational drugs or participated in any clinical study within 60 days or 5 half-lives (if known) of the investigational drug's PK, PD, or biological activity (if known), whichever is longer, prior to administration of the first dose of study drug in this study or is currently participating in another clinical study.
* Prior exposure to exenatide (Byetta® or Bydureon®).
* Significant blood loss (> 450 mL) or has donated 1 or more units of blood or plasma within 6 weeks prior to study randomization.
* History of hypoglycemia.
* History of gastroparesis.
* History of pancreatitis.
* Positive urine results for drugs of abuse, alcohol, or cotinine screen.
* Positive screen for HIV-1 and HIV-2 antibodies, HBsAg, or HCV antibody.
* Clinically significant cardiac changes demonstrated by ECG at screening or Day-1 including:

  * QTcF interval > 450 msec
  * PR interval ≤ 110 msec or > 240 msec
  * Evidence of second- or third-degree atrioventricular block
  * Pathological Q-waves (defined as Q-wave > 40 msec or depth greater than 0.5 mV)
  * Evidence of ventricular pre-excitation
  * Evidence of complete left BBB, incomplete left BBB, complete right BBB
  * Intraventricular conduction delay with QRS duration > 120 msec
  * Bradycardia (defined as sinus rate < 50 bpm) or tachycardia (defined as sinus rate > 100 bpm)
* Has any of the following abnormal vital signs at screening or Day-1:

  * Pulse < 40 or > 100 bpm
  * Respiratory rate < 8 or > 20 breaths per minute
  * Systolic blood pressure < 95 or > 145 mmHg
  * Diastolic blood pressure < 45 or > 90 mmHg
* Serum potassium, chloride, calcium, or sodium outside the normal reference range at screening
* Hepatic transaminases (ALT or AST) > 100 IU/mL at screening.
* Any hematology, chemistry, or urinalysis test results that are clinically significant.
* Any other condition or prior therapy that, in the investigator's opinion, would make the subject unsuitable for the study, or unable or unwilling to comply with the study procedures.
* Unwilling or unlikely to comply with the requirements of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Treatment-Related Adverse Events | Day 1 through Day 29 (Part A) or Day 57 (Part B)
  Frequency and intensity of treatment-related adverse events as assessed using the CTCAE v4.03 criteria and the DMID Adult Toxicity Table for GI-related events.

SECONDARY OUTCOMES:
Pharmacokinetics of NLY01 | Periodic, predose through Day 29 (Part A) or Day 57 (Part B)
  Serum concentration-time profiles for NLY01
Immunogenicity | Periodic, predose through Day 29 (Part A) or Day 57 (Part B)
  Serum anti-drug antibody assessment

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel DeNoia, MD, Principal Investigator — ICON Early Phase Services/CRU
Locations (1):
- ICON Early Phase Services/CRU, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
As a Phase 1 safety study, data will be limited to adverse events and PK. This data will be provided in summary form and/or with descriptive statistics. Individual listings are not expected to provide further insight.

REFERENCES:
- [Background] Yun SP, Kam TI, Panicker N, Kim S, Oh Y, Park JS, Kwon SH, Park YJ, Karuppagounder SS, Park H, Kim S, Oh N, Kim NA, Lee S, Brahmachari S, Mao X, Lee JH, Kumar M, An D, Kang SU, Lee Y, Lee KC, Na DH, Kim D, Lee SH, Roschke VV, Liddelow SA, Mari Z, Barres BA, Dawson VL, Lee S, Dawson TM, Ko HS. Block of A1 astrocyte conversion by microglia is neuroprotective in models of Parkinson's disease. Nat Med. 2018 Jul;24(7):931-938. doi: 10.1038/s41591-018-0051-5. Epub 2018 Jun 11. PMID 29892066
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581
- See also: Neuraly, Inc website — http://www.neuralymed.com
- See also: ICON Early Phase Services - Clinical Trial Site — https://study-volunteers.iconplc.com/study-volunteers/